CLINICAL TRIAL: NCT01953692
Title: A Phase Ib Multi-Cohort Trial of MK-3475 (Pembrolizumab) in Subjects With Hematologic Malignancies
Brief Title: A Trial of Pembrolizumab (MK-3475) in Participants With Blood Cancers (MK-3475-013/KEYNOTE-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-013; 2013-001603-37 (EudraCT Number); MK-3475-013 (Other: Merck)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Myelodysplastic Syndrome; Multiple Myeloma; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Primary Mediastinal B-Cell Lymphoma
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Myelodysplastic Syndromes; Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — pembrolizumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: Myelodysplastic Syndrome (MDS) (Experimental): Participants received pembrolizumab 10 mg/kg by intravenous (IV) infusion on Day 1 of each 14-day cycle.
  Interventions: Biological: Pembrolizumab
- Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM) (Experimental): Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle OR 10 mg/kg by intravenous (IV) infusion on Day 1 of each 14-day cycle.
  Interventions: Biological: Pembrolizumab
- Cohort 3: Relapsed/Refractory (R/R) Hodgkin lymphoma (HL) (Experimental): Participants received pembrolizumab 10 mg/kg by intravenous (IV) infusion on Day 1 of each 14-day cycle.
  Interventions: Biological: Pembrolizumab
- Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) (Experimental): Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle OR 10 mg/kg by intravenous (IV) infusion on Day 1 of each 14-day cycle.
  Interventions: Biological: Pembrolizumab
- Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas (Experimental): Participants received pembrolizumab 10 mg/kg by intravenous (IV) infusion on Day 1 of each 14-day cycle.
  Interventions: Biological: Pembrolizumab
- Cohort 4C: R/R Follicular Lymphoma (FL) (Experimental): Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Pembrolizumab
- Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) (Experimental): Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Pembrolizumab
- Cohort 5: R/R DLBCL pembrolizumab+lenalidomide 20 mg (Experimental): Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle + lenalidomide 20 mg orally (PO) every day (QD) for 21 consecutive days with 7 days off within 28-day cycles.
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide 20 mg
- Cohort 5: R/R DLBCL pembrolizumab+lenalidomide 25 mg (Experimental): Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle + lenalidomide 25 mg PO QD for 21 consecutive days with 7 days off within 28-day cycles.
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide 25 mg

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenalidomide 20 mg — oral capsule
  Other Names: REVLIMID®
  Arms: Cohort 5: R/R DLBCL pembrolizumab+lenalidomide 20 mg
Drug: Lenalidomide 25 mg — oral capsule
  Other Names: REVLIMID®
  Arms: Cohort 5: R/R DLBCL pembrolizumab+lenalidomide 25 mg

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, and efficacy of pembrolizumab (MK-3475, KEYTRUDA®) and pembrolizumab in combination with lenalidomide (Cohort 5 only) in hematologic malignancies. The primary study hypotheses are that treatment with pembrolizumab will result in a clinically meaningful improvement in Objective Response Rate (ORR) or Complete Remission Rate (CRR).

The study includes an initial dose determination to establish the recommended phase 2 dose (RP2D) of lenalidomide given in combination with pembrolizumab in Cohort 5.

With Protocol Amendment 08, enrollment in the Multiple Myeloma arm (Cohort 2) has been completed and no further enrollment will be allowed and enrollment in the Non-Hodgkin Lymphoma Diffuse Large B Cell Lymphoma arm (Cohort 5) has been discontinued and no further enrollment will be allowed.

ELIGIBILITY:
Inclusion criteria:

* Has confirmed diagnosis of relapse or refractory Multiple Myeloma (enrollment completed), Primary mediastinal Large B cell Lymphoma, non-Hodgkin lymphoma (NHL), Follicular Lymphoma, Diffuse Large B cell lymphoma (enrollment discontinued), Hodgkin lymphoma or Myelodysplastic syndrome (enrollment completed).
* Has measurable disease
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Demonstrates adequate organ function
* Prior therapy criteria must be met
* Female participants of childbearing potential and male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Female participants of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study therapy

Exclusion Criteria:

* Is currently participating in and receiving study therapy or has participated in a study of an investigational agent or used an investigational device within 4 weeks of the first dose of study therapy
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years, has received a live vaccine within 30 days of planned start of study therapy, has received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1, received a monoclonal antibody within 4 weeks prior to study Day 1 or has not recovered from adverse events due to a previously administered agent
* Has known clinically active central nervous system (CNS) involvement
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has evidence of interstitial lung disease, active non-infectious pneumonitis, a known additional malignancy that is progressing or requires active treatment, an active infection requiring intravenous systemic therapy, an active autoimmune disease that has required systemic therapy, a known Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV) infection
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study starting with the pre-screening or screening visit through 120 days after the last dose of study therapy
* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has known symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Armand P, Shipp MA, Ribrag V, Michot JM, Zinzani PL, Kuruvilla J, Snyder ES, Ricart AD, Balakumaran A, Rose S, Moskowitz CH. Programmed Death-1 Blockade With Pembrolizumab in Patients With Classical Hodgkin Lymphoma After Brentuximab Vedotin Failure. J Clin Oncol. 2016 Nov 1;34(31):3733-3739. doi: 10.1200/JCO.2016.67.3467. PMID 27354476
- [Result] Ribrag V, Avigan DE, Green DJ, Wise-Draper T, Posada JG, Vij R, Zhu Y, Farooqui MZH, Marinello P, Siegel DS. Phase 1b trial of pembrolizumab monotherapy for relapsed/refractory multiple myeloma: KEYNOTE-013. Br J Haematol. 2019 Aug;186(3):e41-e44. doi: 10.1111/bjh.15888. Epub 2019 Apr 1. No abstract available. PMID 30937889
- [Derived] Kuruvilla J, Armand P, Hamadani M, Kline J, Moskowitz CH, Avigan D, Brody JD, Ribrag V, Herrera AF, Morschhauser F, Kanate A, Zinzani PL, Bitran J, Ghesquieres H, Schuster SJ, Farooqui M, Marinello P, Bartlett NL. Pembrolizumab for patients with non-Hodgkin lymphoma: phase 1b KEYNOTE-013 study. Leuk Lymphoma. 2023 Jan;64(1):130-139. doi: 10.1080/10428194.2022.2136956. Epub 2022 Nov 18. PMID 36398795
- [Derived] Garcia-Manero G, Ribrag V, Zhang Y, Farooqui M, Marinello P, Smith BD. Pembrolizumab for myelodysplastic syndromes after failure of hypomethylating agents in the phase 1b KEYNOTE-013 study. Leuk Lymphoma. 2022 Jul;63(7):1660-1668. doi: 10.1080/10428194.2022.2034155. Epub 2022 Mar 4. PMID 35244520
- [Derived] Griffin GK, Weirather JL, Roemer MGM, Lipschitz M, Kelley A, Chen PH, Gusenleitner D, Jeter E, Pak C, Gjini E, Chapuy B, Rosenthal MH, Xu J, Chen BJ, Sohani AR, Lovitch SB, Abramson JS, Ishizuka JJ, Kim AI, Jacobson CA, LaCasce AS, Fletcher CD, Neuberg D, Freeman GJ, Hodi FS, Wright K, Ligon AH, Jacobsen ED, Armand P, Shipp MA, Rodig SJ. Spatial signatures identify immune escape via PD-1 as a defining feature of T-cell/histiocyte-rich large B-cell lymphoma. Blood. 2021 Mar 11;137(10):1353-1364. doi: 10.1182/blood.2020006464. PMID 32871584
- [Derived] Armand P, Kuruvilla J, Michot JM, Ribrag V, Zinzani PL, Zhu Y, Marinello P, Nahar A, Moskowitz CH. KEYNOTE-013 4-year follow-up of pembrolizumab in classical Hodgkin lymphoma after brentuximab vedotin failure. Blood Adv. 2020 Jun 23;4(12):2617-2622. doi: 10.1182/bloodadvances.2019001367. PMID 32556281
- [Derived] Armand P, Rodig S, Melnichenko V, Thieblemont C, Bouabdallah K, Tumyan G, Ozcan M, Portino S, Fogliatto L, Caballero MD, Walewski J, Gulbas Z, Ribrag V, Christian B, Perini GF, Salles G, Svoboda J, Zain J, Patel S, Chen PH, Ligon AH, Ouyang J, Neuberg D, Redd R, Chatterjee A, Balakumaran A, Orlowski R, Shipp M, Zinzani PL. Pembrolizumab in Relapsed or Refractory Primary Mediastinal Large B-Cell Lymphoma. J Clin Oncol. 2019 Dec 1;37(34):3291-3299. doi: 10.1200/JCO.19.01389. Epub 2019 Oct 14. PMID 31609651
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Zinzani PL, Ribrag V, Moskowitz CH, Michot JM, Kuruvilla J, Balakumaran A, Zhang Y, Chlosta S, Shipp MA, Armand P. Safety and tolerability of pembrolizumab in patients with relapsed/refractory primary mediastinal large B-cell lymphoma. Blood. 2017 Jul 20;130(3):267-270. doi: 10.1182/blood-2016-12-758383. Epub 2017 May 10. PMID 28490569
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included an initial dose determination for Cohort 5 to determine the recommended Phase 2 dose (RP2D) of lenalidomide. Participants started at a dose of 25 mg. The RP2D dose was set at 20 mg and subsequent participants were enrolled at that dose.
Pre-assignment Details: Participants were enrolled in disease-specific cohorts (C): C1: myelodysplastic syndrome (MDS); C2: multiple myeloma (MM); C3: Hodgkin lymphoma (HL); C4: non-Hodgkin lymphoma consisting of:
  * 4A: primary mediastinal B-cell lymphoma (PMBCL)
  * 4B: Non-PMBCL + programmed cell death ligand 1 positive. DLBCL and FL were included in 4C and 4D. The remaining diseases in 4B were classified as "Other"
  * 4C: follicular lymphoma (FL)
  * 4D: diffuse large B-cell lymphoma (DLBCL) And C5: DLBCL
Groups:
- Cohort 2: Relapsed Refractory or Refractory(rR/R) Multiple Myeloma (MM); Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL): Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle OR 10 mg/kg by IV infusion on Day 1 of each 14-day cycle.
- Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL); Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas: Participants received pembrolizumab 10 mg/kg by IV infusion on Day 1 of each 14-day cycle.
- Cohort 4C: R/R Follicular Lymphoma (FL); Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL): Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle.
- Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D): Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle + lenalidomide 20 mg orally (PO) every day (QD) for 21 consecutive days with 7 days off within 28-day cycles. The 20 mg dose of lenalidomide is the RP2D.
- Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg: Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle + lenalidomide 25 mg PO QD for 21 consecutive days with 7 days off within 28-day cycles. The 25 mg dose of lenalidomide was the starting dose for dose determination.
Period: Overall Study
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS) | Cohort 2: Relapsed Refractory or Refractory(rR/R) Multiple Myeloma (MM) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg
Started | 28 | 30 | 31 | 21 | 4 | 22 | 42 | 13 | 6
Completed | 1 | 5 | 11 | 7 | 1 | 4 | 10 | 3 | 1
Not Completed | 27 | 25 | 20 | 14 | 3 | 18 | 32 | 10 | 5
Not completed — Adverse Event | 5 | 2 | 4 | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 15 | 7 | 5 | 0 | 7 | 20 | 3 | 3
Not completed — Death | 5 | 0 | 2 | 2 | 1 | 3 | 6 | 2 | 1
Not completed — Excluded Medication | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 11 | 4 | 2 | 2 | 1 | 2 | 4 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study for Cohort 5 Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 2 | 0 | 3 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS) | Cohort 2: Relapsed Refractory or Refractory(rR/R) Multiple Myeloma (MM) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg | Total
Number analyzed (Participants) | 28 | 30 | 31 | 21 | 4 | 22 | 42 | 13 | 6 | 197
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.4 (10.4) | 67.9 (7.3) | 34.4 (12.1) | 35.2 (12.0) | 49.3 (10.9) | 62.1 (9.2) | 63.8 (11.5) | 62.6 (13.3) | 65.2 (8.4) | 57.3 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 13 | 14 | 0 | 9 | 16 | 5 | 3 | 83
  Male | 18 | 17 | 18 | 7 | 4 | 13 | 26 | 8 | 3 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 8
  Not Hispanic or Latino | 26 | 18 | 25 | 15 | 3 | 21 | 40 | 10 | 6 | 164
  Unknown or Not Reported | 1 | 12 | 4 | 5 | 1 | 0 | 1 | 1 | 0 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 10
  White | 27 | 25 | 29 | 20 | 4 | 19 | 35 | 12 | 5 | 176
  More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs):
Description: An adverse event was defined as any untoward medical occurrence in a participant administered study treatment and did not necessarily have a causal relationship with this treatment. An adverse event could be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the use of the study treatment was also an adverse event.
Time Frame: Up to approximately 78.5 months
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM); Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL): Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle OR 10 mg/kg by IV infusion on Day 1 of each 14-day cycle.
- Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg: Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle + lenalidomide 25 mg PO QD for 21 consecutive days with 7 days off within 28-day cycles.
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS) | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg
Number analyzed (Participants) | 28 | 30 | 31 | 21 | 4 | 22 | 42 | 13 | 6
Participants | 27 | 28 | 31 | 21 | 4 | 21 | 38 | 13 | 5

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: as for outcome 1
Time Frame: Up to approximately 78.5 months
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS) | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg
Number analyzed (Participants) | 28 | 30 | 31 | 21 | 4 | 22 | 42 | 13 | 6
Participants | 6 | 2 | 3 | 1 | 1 | 3 | 2 | 0 | 1

3. Primary Outcome: Objective Response Rate (ORR) in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. CR was demonstrated by ≤5% myeloblasts with normal maturation of all cell lines in the bone marrow (persistent dysplasia will be noted) and normal findings for hemoglobin, platelet count, neutrophil count, and absence of blasts in the blood. PR was all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pre-treatment but still >5%. Cellularity and morphology are not relevant. Cohort 1 was evaluated statistically by comparing the ORR for pembrolizumab to a fixed efficacy target of 10% using a binomial exact test. The percentage of participants with CR and PR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 27
Percentage of participants | 0.0 [0.0 to 10.5]
Statistical Analysis 1: Comparison: Cohort 1: Myelodysplastic Syndrome (MDS); Comparison to a fixed efficacy target of 10%. H0: p ≤ 0.10 versus H1: p > 0.10; Test type: Superiority; p > 0.9999, exact binomial distribution — one-sided p value

4. Primary Outcome: Objective Response Rate (ORR) in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: ORR was defined as the percentage of the participants with either a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) 2006 response criteria. CR=negative immunofixation of serum and urine+disappearance of soft tissue plasmacytomas+≤5% plasma cells in the bone marrow (BM); sCR=stringent complete response, CR as above+normal serum free light-chain ratio and absence of clonal cells in BM; VGPR=serum+urine M-protein (M-p) by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-p+urine M-p <100 mg/24 hr; PR=≥50% reduction of serum M-p+reduction in 24-hour urine M-p by ≥90% or to <200 mg/24 hours. Cohort 2 was evaluated statistically by comparing the ORR for pembrolizumab to a fixed efficacy target of 25% using a binomial exact test. The percentage of participants with CR, sCR, PR, VGPR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 30
Percentage of participants | 0.0 [0.0 to 9.5]
Statistical Analysis 1: Comparison: Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM); Comparison to a fixed efficacy target of 25%. H0: p ≤ 0.25 versus H1: p > 0.25; Test type: Superiority; p > 0.9999, exact binomial distribution — one-sided p-value

5. Primary Outcome: Complete Remission Rate (CRR) in Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Description: CRR was defined as the percentage of participants with complete remission according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. Complete remission was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. Cohort 3 was evaluated statistically by comparing the complete remission for pembrolizumab to a fixed efficacy target of 10% using a binomial exact test. The percentage of participants with complete remission as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 3 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Number analyzed (Participants) | 31
Percentage of participants | 22.6 [11.1 to 38.3]
Statistical Analysis 1: Comparison: Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL); Comparison to a fixed efficacy target of 10%. H0: p ≤ 0.10 versus H1: p > 0.10; Test type: Superiority; p = 0.0306, exact binomial distribution — one-sided p-value

6. Primary Outcome: Objective Response Rate (ORR) in Participants Pooled From the Cohort 4 Non-Hodgkin Lymphoma (NHL) Sub-Cohorts (Cohorts 4A+4B+4C+4D)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. The pooled Cohort 4 sub-cohorts were evaluated statistically by comparing the ORR for pembrolizumab to a fixed efficacy target of 25% using a binomial exact test. The percentage of participants with CR and PR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from the Cohort 4 NHL sub-cohorts (Cohorts 4A+4B+4C+4D) with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of participants grouped by disease cohort (NHL).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D): Participants from the pooled Cohort 4 NHL sub-cohorts (Cohorts 4A+4B+4C+4D) received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle OR 10 mg/kg by IV infusion on Day 1 of each 14-day cycle.
Arm/Group | Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D)
Number analyzed (Participants) | 86
Percentage of participants | 22.1 [15.0 to 30.7]
Statistical Analysis 1: Comparison: Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D); Comparison to a fixed efficacy target of 25%. H0: p ≤ 0.25 versus H1: p > 0.25; Test type: Superiority; p = 0.7696, exact binomial distribution — one-sided p-value

7. Primary Outcome: Objective Response Rate (ORR) in the Cohort 4 Non-Hodgkin Lymphoma (NHL) Individual Sub-Cohorts (Cohorts 4A, 4B, 4C, and 4D)
Description: ORR was evaluated for each of the Cohort 4 sub-cohorts: 4A (primary mediastinal B-cell lymphoma), 4B (grey zone, splenic marginal zone, and mantle cell lymphomas), 4C (follicular lymphoma), and 4D (diffuse large B-Cell lymphoma). ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. Per protocol, Cohorts 4A, 4B, 4C, and 4D were not planned to be compared to an efficacy target. The percentage of participants with CR and PR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohorts 4A, 4B, 4C, and 4D with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of participants grouped by disease cohort (NHL).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 21 | 4 | 20 | 41
Percentage of participants | 47.6 [28.6 to 67.2] | 50.0 [9.8 to 90.2] | 10.0 [1.8 to 28.3] | 12.2 [4.9 to 23.9]

8. Primary Outcome: Objective Response Rate (ORR) in Participants Pooled From Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide) Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. Per protocol, pooled Cohort 5 was not planned to be evaluated statistically compared to a fixed efficacy target. The percentage of participants with CR and PR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from Cohort 5 (pembrolizumab + 20 or 25 mg doses of lenalidomide) with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (DLBCL) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide): Participants from the pooled Cohort 5 received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle + lenalidomide 20 mg or 25 mg PO QD for 21 consecutive days with 7 days off within 28-day cycles.
Arm/Group | Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide)
Number analyzed (Participants) | 18
Percentage of participants | 38.9 [19.9 to 60.8]

9. Secondary Outcome: Objective Response Rate (ORR) in Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. The percentage of participants who experience ORR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 3 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Number analyzed (Participants) | 31
Percentage of participants | 64.5 [48.2 to 78.7]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study treatment to death due to any cause. OS was calculated from product-limit (Kaplan-Meier) method for censored data. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Time Frame: Up to approximately 78.5 months
Population: All participants with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS) | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 27 | 30 | 31 | 21 | 4 | 20 | 41
Months | 6.0 [3.5 to 12.2] | 20.2 [14.1 to 35.5] | NA [NA to NA] — NA=Median OS and upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event. | 37.1 [4.9 to NA] — NA=OS upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 23.8 [0.4 to 28.6] | NA [14.7 to NA] — NA=Median OS and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 4.9 [3.6 to 7.8]

11. Secondary Outcome: Overall Survival (OS) in Participants Pooled From the Cohort 4 Non-Hodgkin Lymphoma (NHL) Sub-Cohorts (Cohorts 4A+4B+4C+4D)
Description: as for outcome 10
Time Frame: Up to approximately 78.5 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D)
Number analyzed (Participants) | 86
Months | 12.0 [6.0 to 22.5]

12. Secondary Outcome: Overall Survival (OS) in Participants Pooled From Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide) Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Description: as for outcome 10
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from the Cohort 5 (pembrolizumab + 20 or 25 mg doses of lenalidomide) with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (DLBCL) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide)
Number analyzed (Participants) | 18
Months | 23.0 [6.1 to NA] — NA=OS upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

13. Secondary Outcome: Duration of Response (DOR) in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: For participants who demonstrated a confirmed Complete Response (CR) or partial response (PR), DOR was defined as the time from CR or PR to documented disease progression or death. CR and PR were assessed according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. CR was demonstrated by ≤5% myeloblasts with normal maturation of all cell lines in the bone marrow (persistent dysplasia will be noted) and normal findings for hemoglobin, platelet count, neutrophil count, and absence of blasts in the blood. PR was all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pre-treatment but still >5%. Cellularity and morphology are not relevant. DOR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation, at least 1 post-baseline efficacy evaluation, and who demonstrated a PR or CR. DOR was not analyzed because there were no participants who demonstrated a PR or CR in Cohort 1.
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 0

14. Secondary Outcome: Duration of Response (DOR) in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: For participants who demonstrated a confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), DOR was defined as the time from sCR, CR, VGPR, or PR to documented disease progression or death. Response was assessed according to the International Myeloma Working Group (IMWG) 2006 response criteria. CR=negative immunofixation of serum and urine+disappearance of soft tissue plasmacytomas+≤5% plasma cells in the bone marrow (BM); sCR=stringent complete response, CR as above+normal serum free light-chain ratio and absence of clonal cells in BM; VGPR=serum+urine M-protein (M-p) by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-p+urine M-p <100 mg/24 hr; PR=≥50% reduction of serum M-p+reduction in 24-hour urine M-p by ≥90% or to <200 mg/24 hours. DOR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2 with a baseline efficacy evaluation, at least 1 post-baseline efficacy evaluation, and who demonstrated a VGPR, PR, sCR, or CR. DOR was not analyzed because there were no participants who demonstrated a VGPR, PR, sCR, or CR in Cohort 2.
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 0

15. Secondary Outcome: Duration of Response (DOR) in Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Description: For participants who demonstrated a confirmed Complete Response (CR) or partial response (PR), DOR was defined as the time from CR or PR to documented disease progression or death. CR and PR were assessed according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. DOR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 3 with a baseline efficacy evaluation, at least 1 post-baseline efficacy evaluation, and who demonstrated a PR or CR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Number analyzed (Participants) | 20
Months | 25.0 [5.6 to NA] — NA=DOR upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

16. Secondary Outcome: Duration of Response (DOR) in Participants Pooled From the Cohort 4 Non-Hodgkin Lymphoma (NHL) Sub-Cohorts (Cohorts 4A+4B+4C+4D)
Description: as for outcome 15
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from the Cohort 4 NHL sub-cohorts (Cohorts 4A+4B+4C+4D) with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation and who demonstrated a PR or CR. The analysis was pre-specified to be a pooled analysis of participants grouped by disease cohort (NHL).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D)
Number analyzed (Participants) | 19
Months | NA [9.6 to NA] — NA=Median DOR and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

17. Secondary Outcome: Duration of Response (DOR) in the Cohort 4 Non-Hodgkin Lymphoma (NHL) Individual Sub-Cohorts (Cohorts 4A, 4B, 4C, and 4D)
Description: DOR was evaluated for each of the Cohort 4 sub-cohorts: 4A (primary mediastinal B-cell lymphoma), 4B (grey zone, splenic marginal zone, and mantle cell lymphomas), 4C (follicular lymphoma), and 4D (diffuse large B-Cell lymphoma). For participants who demonstrated a confirmed Complete Response (CR) or partial response (PR), DOR was defined as the time from CR or PR to documented disease progression or death. CR and PR were assessed according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. DOR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohorts 4A, 4B, 4C, and 4D with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation and who demonstrated a PR or CR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 10 | 2 | 2 | 5
Months | NA [6.9 to NA] — NA=Median DOR and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [1.7 to NA] — NA=Median DOR and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [NA to NA] — NA=Median DOR and upper and lower limits not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 13.6 [2.6 to NA] — NA=DOR upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

18. Secondary Outcome: Duration of Response (DOR) in Participants Pooled From Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide) Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Description: as for outcome 15
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from the Cohort 5 (pembrolizumab + 20 or 25 mg doses of lenalidomide) with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation and who demonstrated a PR or CR. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (DLBCL) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide)
Number analyzed (Participants) | 7
Months | NA [2.8 to NA] — NA=Median DOR and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

19. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. CR was demonstrated by ≤5% myeloblasts with normal maturation of all cell lines in the bone marrow (persistent dysplasia will be noted) and normal findings for hemoglobin, platelet count, neutrophil count, and absence of blasts in the blood. PR was all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pre-treatment but still >5%. Cellularity and morphology are not relevant. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 positive (PD-L1 of ≥1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1, who were PD-L1 positive, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. ORR by PD-L1 status was not analyzed because there were no participants who demonstrated a PR or CR in Cohort 1.
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 0

20. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Negative Participants in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. CR was demonstrated by ≤5% myeloblasts with normal maturation of all cell lines in the bone marrow (persistent dysplasia will be noted) and normal findings for hemoglobin, platelet count, neutrophil count, and absence of blasts in the blood. PR was all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pre-treatment but still >5%. Cellularity and morphology are not relevant. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 negative (PD-L1 of <1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1, who were PD-L1 negative, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. ORR by PD-L1 status was not analyzed because there were no participants who demonstrated a PR or CR in Cohort 1.
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 0

21. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Indeterminate Participants in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. CR was demonstrated by ≤5% myeloblasts with normal maturation of all cell lines in the bone marrow (persistent dysplasia will be noted) and normal findings for hemoglobin, platelet count, neutrophil count, and absence of blasts in the blood. PR was all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pre-treatment but still >5%. Cellularity and morphology are not relevant. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for participants with an indeterminate (missing) PD-L1 status.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1, who had an indeterminate PD-L1 status, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. ORR by PD-L1 status was not analyzed because there were no participants who demonstrated a PR or CR in Cohort 1.
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 0

22. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: ORR was defined as the percentage of the participants with either a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) 2006 response criteria. CR=negative immunofixation of serum and urine+disappearance of soft tissue plasmacytomas+≤5% plasma cells in the bone marrow (BM); sCR=stringent complete response, CR as above+normal serum free light-chain ratio and absence of clonal cells in BM; VGPR=serum+urine M-protein (M-p) by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-p+urine M-p <100 mg/24 hr; PR=≥50% reduction of serum M-p+reduction in 24-hour urine M-p by ≥90% or to <200 mg/24 hours. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR, sCR, PR, VGPR as assessed by the investigator is presented for PD-L1 positive (PD-L1 of ≥1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2, who were PD-L1 positive, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. ORR by PD-L1 status was not analyzed because there were no participants who demonstrated a PR or CR in Cohort 2.
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 0

23. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Negative Participants in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: ORR was defined as the percentage of the participants with either a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) 2006 response criteria. CR=negative immunofixation of serum and urine+disappearance of soft tissue plasmacytomas+≤5% plasma cells in the bone marrow (BM); sCR=stringent complete response, CR as above+normal serum free light-chain ratio and absence of clonal cells in BM; VGPR=serum+urine M-protein (M-p) by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-p+urine M-p <100 mg/24 hr; PR=≥50% reduction of serum M-p+reduction in 24-hour urine M-p by ≥90% or to <200 mg/24 hours. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR, sCR, PR, VGPR as assessed by the investigator is presented for PD-L1 negative (PD-L1 of <1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2, who were PD-L1 negative, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. ORR by PD-L1 status was not analyzed because there were no participants who demonstrated a PR or CR in Cohort 2.
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 0

24. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Indeterminate Participants in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: ORR was defined as the percentage of the participants with either a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) 2006 response criteria. CR=negative immunofixation of serum and urine+disappearance of soft tissue plasmacytomas+≤5% plasma cells in the bone marrow (BM); sCR=stringent complete response, CR as above+normal serum free light-chain ratio and absence of clonal cells in BM; VGPR=serum+urine M-protein (M-p) by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-p+urine M-p <100 mg/24 hr; PR=≥50% reduction of serum M-p+reduction in 24-hour urine M-p by ≥90% or to <200 mg/24 hours. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR, sCR, PR, VGPR as assessed by the investigator is presented for participants with an indeterminate (missing) PD-L1 status.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2, who had an indeterminate PD-L1 status, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. ORR by PD-L1 status was not analyzed because there were no participants who demonstrated a PR or CR in Cohort 2.
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 0

25. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants in Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 positive (PD-L1 of ≥1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 3, who were PD-L1 positive, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Number analyzed (Participants) | 11
Percentage of participants | 54.5 [23.4 to 83.3]

26. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Negative Participants in Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 negative (PD-L1 of <1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 3, who were PD-L1 negative, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Number analyzed (Participants) | 2
Percentage of participants | 50.0 [1.3 to 98.7]

27. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Indeterminate Participants in Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for participants with an indeterminate (missing) PD-L1 status.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 3, who had an indeterminate PD-L1 status, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Number analyzed (Participants) | 18
Percentage of participants | 72.2 [46.5 to 90.3]

28. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants Pooled From the Cohort 4 Non-Hodgkin Lymphoma (NHL) Sub-Cohorts (Cohorts 4A+4B+4C+4D)
Description: as for outcome 25
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from the Cohort 4 NHL sub-cohorts (Cohorts 4A+4B+4C+4D), who were PD-L1 positive, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of participants grouped by disease cohort (NHL).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D)
Number analyzed (Participants) | 32
Percentage of participants | 18.8 [7.2 to 36.4]

29. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Negative Participants Pooled From the Cohort 4 Non-Hodgkin Lymphoma (NHL) Sub-Cohorts (Cohorts 4A+4B+4C+4D)
Description: as for outcome 26
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from the Cohort 4 NHL sub-cohorts (Cohorts 4A+4B+4C+4D), who were PD-L1 negative, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of participants grouped by disease cohort (NHL).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D)
Number analyzed (Participants) | 35
Percentage of participants | 11.4 [3.2 to 26.7]

30. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Indeterminate Participants Pooled From the Cohort 4 Non-Hodgkin Lymphoma (NHL) Sub-Cohorts (Cohorts 4A+4B+4C+4D)
Description: as for outcome 27
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from the Cohort 4 NHL sub-cohorts (Cohorts 4A+4B+4C+4D), who had an indeterminate PD-L1 status, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of participants grouped by disease cohort (NHL).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D)
Number analyzed (Participants) | 19
Percentage of participants | 47.4 [24.4 to 71.1]

31. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants in the Cohort 4 Non-Hodgkin Lymphoma (NHL) Individual Sub-Cohorts (Cohorts 4A, 4B, 4C, and 4D)
Description: ORR was evaluated for each of the Cohort 4 sub-cohorts: 4A (primary mediastinal B-cell lymphoma), 4B (grey zone, splenic marginal zone, and mantle cell lymphomas), 4C (follicular lymphoma), and 4D (diffuse large B-Cell lymphoma). ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 positive (PD-L1 of ≥1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohorts 4A, 4B, 4C, and 4D, who were PD-L1 positive, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 11 | 2 | 4 | 15
Percentage of participants | 27.3 [6.0 to 61.0] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 60.2] | 6.7 [0.2 to 31.9]

32. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Negative Participants in the Cohort 4 Non-Hodgkin Lymphoma (NHL) Individual Sub-Cohorts (Cohorts 4A, 4B, 4C, and 4D)
Description: ORR was evaluated for each of the Cohort 4 sub-cohorts: 4A (primary mediastinal B-cell lymphoma), 4B (grey zone, splenic marginal zone, and mantle cell lymphomas), 4C (follicular lymphoma), and 4D (diffuse large B-Cell lymphoma). ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 negative (PD-L1 of <1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohorts 4A, 4B, 4C, and 4D, who were PD-L1 negative, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 4 | 2 | 14 | 15
Percentage of participants | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 84.2] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8]

33. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Indeterminate Participants in the Cohort 4 Non-Hodgkin Lymphoma (NHL) Individual Sub-Cohorts (Cohorts 4A, 4B, 4C, and 4D)
Description: ORR was evaluated for each of Cohort 4 sub-cohorts: 4A (primary mediastinal B-cell lymphoma), 4B (grey zone, splenic marginal zone, and mantle cell lymphomas), 4C (follicular lymphoma), and 4D (diffuse large B-Cell lymphoma). ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in bone marrow, spleen, liver, and lymph nodes. PR was >50% decrease in the sum of product diameters (SPD) for ≤6 target masses for lymph nodes and >50% decrease in SPD for a single nodule in greatest transverse diameter for spleen and liver, and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for participants with an indeterminate (missing) PD-L1 status.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohorts 4A, 4B, 4C, and 4D, who had an indeterminate PD-L1 status, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. ORR was not analyzed for Cohort 4B because there were no participants with a PD-L1 status of indeterminate in this Cohort.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 6 | 0 | 2 | 11
Percentage of participants | 66.7 [22.3 to 95.7] |  | 50.0 [1.3 to 98.7] | 36.4 [10.9 to 69.2]

34. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants Pooled From Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide): Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and for nodal masses. PR was >50% decrease in the sum of product diameters for ≤6 target dominant masses for lymph nodes, spleen nodules, and liver nodules and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 positive (PD-L1 of ≥1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from Cohort 5 (pembrolizumab + 20 or 25 mg doses of lenalidomide), who were PD-L1 positive, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (DLBCL) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide)
Number analyzed (Participants) | 4
Percentage of participants | 75.0 [19.4 to 99.4]

35. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Negative Participants Pooled From Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide): Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and for nodal masses. PR was >50% decrease in the sum of product diameters for ≤6 target dominant masses for lymph nodes, spleen nodules, and liver nodules and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for PD-L1 negative (PD-L1 of <1%) participants.
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from Cohort 5 (pembrolizumab + 20 or 25 mg doses of lenalidomide), who were PD-L1 negative, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (DLBCL) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide)
Number analyzed (Participants) | 8
Percentage of participants | 25.0 [3.2 to 65.1]

36. Secondary Outcome: Objective Response Rate (ORR) in Programmed Cell Death Ligand 1 (PD-L1) Indeterminate Participants Pooled From Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide): Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Description: ORR was defined as the percentage of participants with response (complete response [CR] or partial response [PR]) according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. CR was demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and for nodal masses. PR was >50% decrease in the sum of product diameters for ≤6 target dominant masses for lymph nodes, spleen nodules, and liver nodules and no size increase in the lymph nodes, spleen, or liver. PD-L1 was assessed by immunohistochemistry (IHC). The percentage of participants with CR and PR as assessed by the investigator is presented for participants with an indeterminate (missing) PD-L1 status.
Time Frame: Up to approximately 78.5 months
Population: All participants pooled from Cohort 5 (pembrolizumab + 20 or 25 mg doses of lenalidomide), who had an indeterminate PD-L1 status, with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation. The analysis was pre-specified to be a pooled analysis of all participants grouped by disease cohort (DLBCL) and treatment combination (irrespective of dose); therefore data by individual dose were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide)
Number analyzed (Participants) | 6
Percentage of participants | 33.3 [4.3 to 77.7]

37. Secondary Outcome: Progression-free Survival (PFS) in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. PD was assessed according to the International Myeloma Working Group (IMWG) 2006 response criteria. PD was defined as ≥1 of the following: increase of ≥25% from baseline of serum or urine M-component or >10 mg/dl difference between involved and uninvolved free light chain levels; development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; or hypercalcemia. PFS was calculated from the Kaplan-Meier method for censored data. PFS as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 30
Months | 2.7 [1.4 to 13.0]

38. Secondary Outcome: Progression-free Survival (PFS) in Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Description: PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. PD was assessed according to the revised response criteria for malignant lymphoma per Cheson et al. 2007. PD was the appearance of any new lesion, >50% increase in the sum of product diameters (SPD) of ≥1 lymph node, or a >50% increase in the longest diameter of a previous lymph node, lesions positron emission tomography (PET) positive if 18F-fluorodeoxyglucose (FDG)-avid lymphoma or PET positive prior to therapy for lymph nodes; >50% increase from nadir in the SPD of previous lesions in the liver and spleen; or new or recurrent involvement of the bone marrow. PFS was calculated from the Kaplan-Meier method for censored data. PFS as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 3 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL)
Number analyzed (Participants) | 31
Months | 8.7 [4.9 to 28.1]

39. Secondary Outcome: Progression-free Survival (PFS) in Participants Pooled From the Cohort 4 Non-Hodgkin Lymphoma (NHL) Sub-Cohorts (Cohorts 4A+4B+4C+4D)
Description: as for outcome 38
Time Frame: Up to approximately 78.5 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pooled Cohort 4 Sub-cohorts (Cohorts 4A+4B+4C+4D)
Number analyzed (Participants) | 86
Months | 1.7 [1.4 to 2.7]

40. Secondary Outcome: Progression-free Survival (PFS) in the Cohort 4 Non-Hodgkin Lymphoma (NHL) Individual Sub-Cohorts (Cohorts 4A, 4B, 4C, and 4D)
Description: as for outcome 38
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohorts 4A, 4B, 4C, and 4D with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 21 | 4 | 20 | 41
Months | 19.0 [1.9 to NA] — NA=PFS upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 7.3 [0.3 to 10.3] | 1.7 [1.3 to 3.4] | 1.4 [1.3 to 1.7]

41. Secondary Outcome: Progression-free Survival (PFS) in Participants Pooled From the Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide) Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Description: as for outcome 38
Time Frame: Up to approximately 78.5 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pooled Cohort 5 (Pembrolizumab + 20 or 25 mg Doses of Lenalidomide)
Number analyzed (Participants) | 18
Months | 5.5 [2.7 to NA] — NA=PFS upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

42. Secondary Outcome: Marrow Complete Response (mCR) in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: mCR was defined as ≤5% myeloblasts in the bone marrow with a decrease in myeloblasts ≥50% over pretreatment according to the modified International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. The percentage of participants with mCR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 27
Percentage of participants | 18.5 [7.6 to 35.1]

43. Secondary Outcome: Cytogenic Complete Response in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: Cytogenic complete response was evaluated by detection of chromosomal abnormalities by cytogenic techniques and assessed according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. Cytogenic complete response was defined as the disappearance of the chromosomal abnormality detected pre-treatment without the appearance of new chromosomal abnormalities. The percentage of participants with cytogenic complete response as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 27
Percentage of participants | 11.1 [3.1 to 26.3]

44. Secondary Outcome: Cytogenic Partial Response in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: Cytogenic partial response was evaluated by detection of chromosomal abnormalities by cytogenic techniques and assessed according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. Cytogenic partial response was defined as ≥50% reduction of the chromosomal abnormality detected pre-treatment. The percentage of participants with cytogenic partial response as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 27
Percentage of participants | 11.1 [3.1 to 26.3]

45. Secondary Outcome: Erythroid Response in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: Erythroid response was measured as an evaluation of hematologic improvement and was assessed according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. Erythroid response baseline was based on an average of at least 2 pre-treatment measurements taken ≥1 week apart and not influenced by transfusions. Responses were considered significant if they lasted for ≥8 weeks. Criteria for an erythroid response include: hemoglobin (Hgb) increase by ≥1.5 grams/deciliter (g/dl) from pretreatment or reduction of ≥4 transfusions/8 weeks compared with the pre-treatment transfusion number in the previous 8 weeks. Only transfusions given for a Hgb of ≤9.0 g/dl pretreatment counted for response evaluation. The percentage of participants with an erythroid response as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 27
Percentage of participants | 7.1 [1.3 to 21.5]

46. Secondary Outcome: Neutrophil Response in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: Neutrophil response was measured as an evaluation of hematologic improvement and was assessed according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. Neutrophil response baseline was based on an average of at least 2 pre-treatment measurements taken ≥1 week apart and not influenced by transfusions. Responses were considered significant if they lasted for ≥8 weeks. Criterion for a neutrophil response was a ≥100% increase in neutrophil count from pre-treatment and an absolute increase of >0.5 x 10^9/Liter. The percentage of participants with a neutrophil response as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 27
Percentage of participants | 3.6 [0.2 to 16.4]

47. Secondary Outcome: Platelet Response in Cohort 1: Myelodysplastic Syndrome (MDS)
Description: Platelet response was measured as an evaluation of hematologic improvement and was assessed according to the International Working Group (IWG) response criteria in myelodysplasia per Cheson et al. 2006. Platelet response baseline was based on an average of at least 2 pre-treatment measurements taken ≥1 week apart and not influenced by transfusions. Responses were considered significant if they lasted for ≥8 weeks. Criterion for a platelet response was an absolute increase of ≥30 x 10^9/Liter platelet count for participants with a pre-treatment count of ≥20 x 10^9/Liter and for participants with a pre-treatment count of <20 x 10^9/Liter there must have been an absolute increase to ≥20 x 10^9/Liter and a ≥100% increase in pre-treatment level. The percentage of participants with a platelet response as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 1 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 27
Percentage of participants | 7.1 [1.3 to 21.5]

48. Secondary Outcome: Time to Progression (TTP) in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: TTP was defined as the time from first dose of study treatment to disease progression. Progressive disease was assessed according to the International Myeloma Working Group (IMWG) 2006 response criteria. PD was defined as ≥1 of the following: increase of ≥25% from baseline of serum or urine M-component or >10 mg/dl difference between involved and uninvolved free light chain levels; development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; bone marrow plasma cell percentage absolute % must be ≥10%; or hypercalcemia. The TTP as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 30
Months | 2.7 [1.4 to 2.8]

49. Secondary Outcome: Stringent Complete Remission (sCR) in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: sCR was assessed according to the International Myeloma Working Group (IMWG) 2006 response criteria. sCR was defined as complete response [CR] plus normal serum free light-chain ratio and absence of clonal cells in bone marrow. CR criteria are negative immunofixation of serum and urine and disappearance of soft tissue plasmacytomas and ≤5% plasma cells in the bone marrow. The percentage of participants with sCR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of partiicpants
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 30
Percentage of partiicpants | 0.0 [0.0 to 9.5]

50. Secondary Outcome: Complete Response (CR) in Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Description: CR was assessed according to the International Myeloma Working Group (IMWG) 2006 response criteria. CR was defined as negative immunofixation of serum and urine and disappearance of soft tissue plasmacytomas and <5% plasmacytomas in the bone marrow. The percentage of participants with CR as assessed by the investigator is presented.
Time Frame: Up to approximately 78.5 months
Population: All participants in Cohort 2 with a baseline efficacy evaluation and at least 1 post-baseline efficacy evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Relapsed Refractory/Refractory (rR/R) Multiple Myeloma (MM)
Number analyzed (Participants) | 30
Percentage of participants | 0.0 [0.0 to 9.5]

ADVERSE EVENTS:
Time Frame: Up to approximately 78.5 months
Description: The analysis population for adverse events (AEs) consisted of all participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE unless considered related to study treatment. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "neoplasm progression", "malignant neoplasm progression" and "disease progression" not related to study treatment are excluded.
Arm/Group | Cohort 1: Myelodysplastic Syndrome (MDS) | Cohort 2: Relapsed Refractory or Refractory(rR/R) Multiple Myeloma (MM) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas | Cohort 4C: R/R Follicular Lymphoma (FL) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg
All-Cause Mortality (participants affected / at risk) | 25/28 | 23/30 | 8/31 | 11/21 | 4/4 | 11/22 | 37/42 | 8/13 | 4/6
Serious Adverse Events (participants affected / at risk) | 20/28 | 9/30 | 13/31 | 8/21 | 2/4 | 8/22 | 22/42 | 4/13 | 1/6
Other Adverse Events (participants affected / at risk) | 25/28 | 27/30 | 30/31 | 21/21 | 4/4 | 21/22 | 34/42 | 13/13 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Myelodysplastic Syndrome (MDS) (N=28) | Cohort 2: Relapsed Refractory or Refractory(rR/R) Multiple Myeloma (MM) (N=30) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) (N=31) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) (N=21) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas (N=4) | Cohort 4C: R/R Follicular Lymphoma (FL) (N=22) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) (N=42) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D) (N=13) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Myelodysplastic Syndrome (MDS) (N=28) | Cohort 2: Relapsed Refractory or Refractory(rR/R) Multiple Myeloma (MM) (N=30) | Cohort 3: Relapsed/Refractory (R/R) Hodgkin Lymphoma (HL) (N=31) | Cohort 4A: R/R Primary Mediastinal B-cell Lymphoma (PMBCL) (N=21) | Cohort 4B: Other Non-Hodgkin Lymphoma: Grey Zone, Splenic Marginal Zone, and Mantle Cell Lymphomas (N=4) | Cohort 4C: R/R Follicular Lymphoma (FL) (N=22) | Cohort 4D: R/R Diffuse Large B-Cell Lymphoma (DLBCL) (N=42) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 20 mg (RP2D) (N=13) | Cohort 5: R/R DLBCL Pembrolizumab+Lenalidomide 25 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 11 (12) | 6 (6) | 5 (8) | 0 (0) | 4 (4) | 10 (14) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (15) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 4 (15) | 7 (10) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (2) | 0 (0) | 2 (3) | 4 (6) | 3 (4) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 1 (1) | 5 (5) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (4) | 2 (3) | 0 (0) | 4 (5) | 7 (8) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (3) | 8 (11) | 3 (3) | 0 (0) | 3 (4) | 8 (8) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 11 (13) | 7 (10) | 2 (2) | 6 (7) | 6 (6) | 4 (7) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 8 (11) | 5 (6) | 1 (1) | 4 (4) | 12 (12) | 2 (3) | 1 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 2 (3) | 0 (0) | 4 (4) | 7 (9) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 11 (11) | 7 (9) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 2 (4) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 12 (13) | 2 (2) | 6 (7) | 3 (5) | 2 (2) | 10 (11) | 15 (16) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 5 (5) | 6 (6) | 2 (2) | 2 (4)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (6) | 1 (2) | 5 (5) | 6 (8) | 1 (1) | 3 (4) | 7 (8) | 1 (1) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (4) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (4) | 1 (3) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 4 (6) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (8) | 2 (2) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 6 (6) | 5 (5) | 3 (3) | 0 (0) | 3 (4) | 9 (9) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (5) | 2 (3) | 0 (0) | 1 (2) | 8 (13) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (3) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 4 (10) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 4 (12) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 4 (11) | 2 (2) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8) | 4 (5) | 0 (0) | 0 (0) | 6 (7) | 7 (7) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 8 (9) | 4 (5) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 2 (4) | 4 (5) | 1 (1) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (5) | 1 (2) | 2 (3) | 1 (1) | 4 (5) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 12 (19) | 12 (15) | 1 (2) | 4 (4) | 5 (7) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2) | 10 (11) | 2 (2) | 0 (0) | 3 (3) | 6 (6) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (6) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 8 (10) | 3 (4) | 0 (0) | 1 (1) | 5 (6) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 3 (4) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 4 (5) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment of participants into Cohort 5 of this study was discontinued after the Food and Drug Administration (FDA) implemented a clinical hold after determining the risks of pembrolizumab + lenalidomide outweighed any potential benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT01953692/Prot_SAP_000.pdf